CLINICAL TRIAL: NCT03653026
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Induction Study to Evaluate the Efficacy and Safety of Upadacitinib (ABT-494) in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of the Efficacy and Safety of Upadacitinib (ABT-494) in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: U-Accomplish
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-675; 2016-000642-62 (EudraCT Number)
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Results first posted 2021-11-26 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Upadacitinib; ABT-494; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upadacitinib 45 mg (Experimental): Participants received 45 mg upadacitinib once daily (QD) for 8 weeks. Participants who did not achieve clinical response per Adapted Mayo score at Week 8 received upadacitinib 45 mg once daily for 8 additional weeks in the open-label extension period.
  Interventions: Drug: Upadacitinib
- Placebo (Placebo Comparator): Participants received placebo matching to upadacitinib once daily for 8 weeks. Participants who did not achieve clinical response per Adapted Mayo score at Week 8 received upadacitinib 45 mg once daily for 8 weeks in the open-label extension period.
  Interventions: Drug: Placebo; Drug: Upadacitinib

INTERVENTIONS:
Drug: Placebo — Tablet for oral administration
  Arms: Placebo
Drug: Upadacitinib — Tablet for oral administration
  Other Names: ABT-494; RINVOQ®

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of upadacitinib compared to placebo in inducing clinical remission (per Adapted Mayo score) in participants with moderately to severely active ulcerative colitis (UC).

DETAILED DESCRIPTION:
Study M14-675 consists of 2 parts, Part 1 and Part 2. Part 1 is a randomized, double-blind, placebo-controlled 8-week induction period. Part 2 is an open-label, 8-week extended treatment period for participants who did not achieve clinical response at Week 8 in Part 1.

Eligible participants are randomized in a 2:1 ratio to one of the two treatment groups (upadacitinib 45 mg or matching placebo) for 8 weeks. The randomization is stratified by biologic inadequate responder (bio-IR) status (bio-IR vs non-bio-IR), corticosteroid use (yes or no), and Adapted Mayo score (≤ 7 or > 7) at Baseline. Within bio-IR, the randomization is further stratified by number of prior biologic treatments (≤ 1 or > 1). Within non-bio-IR, the randomization is further stratified by previous biologic use (yes or no).

Participants who achieve clinical response defined by Adapted Mayo Score at Week 8 or Week 16 and do not meet any study discontinuation criteria are eligible to enroll into Study M14-234 Substudy 3 (NCT02819635; 52-week maintenance study) or Study M14-533 Cohort 1 (NCT03006068; long-term follow-up study).

ELIGIBILITY:
Inclusion Criteria:

- Male or female participants ≥ 16 and ≤ 75 years of age at Baseline Note: Adolescent participants at the age of 16 or 17 years old will be eligible to participate if approved by the country or regulatory/health authorities.

Note: Adolescent participants at the age of 16 or 17 years old must weigh ≥ 40 kilograms and meet the definition of Tanner Stage 5 at the Screening Visit.

* Diagnosis of Ulcerative Colitis (UC) for 90 days or greater prior to Baseline, confirmed by colonoscopy during the Screening Period, with exclusion of current infection, colonic dysplasia and/or malignancy. Appropriate documentation of biopsy results consistent with the diagnosis of UC, in the assessment of the Investigator, must be available.
* Active UC with an Adapted Mayo score of 5 to 9 points and endoscopic subscore of 2 to 3.
* Demonstrated an inadequate response, loss of response, or intolerance to at lease one of the following treatments including, oral aminosalicylates, corticosteroids, immunosuppressants, and/or biologic therapies.

Note: Participants who have had inadequate response, loss of response to conventional therapy but have not failed biologic therapy (Non-bio-IR) and have received a prior biologic for up to 1 year may be enrolled, however they must have discontinued the biologic for reasons other than inadequate response or intolerance (e.g., change of insurance, well controlled disease), and must meet criteria for inadequate response, loss of response, or intolerance as defined above.

* Female Participants of childbearing potential must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at the Baseline Visit.
* If female, participant must meet the contraception recommendation criteria.

Exclusion Criteria:

* Participant with current diagnosis of Crohn's disease (CD) or diagnosis of indeterminate colitis (IC).
* Current diagnosis of fulminant colitis and/or toxic megacolon.
* Participant with disease limited to the rectum (ulcerative proctitis) during the Screening endoscopy.
* Received cyclosporine, tacrolimus, mycophenolate mofetil, or thalidomide within 30 days prior to Baseline.
* Participant who received azathioprine or 6-mercaptopurine (6-MP) within 10 days of Baseline.
* Received intravenous corticosteroids within 14 days prior to Screening or during the Screening Period.
* Participant with previous exposure to Janus Activated Kinase (JAK) inhibitor (e.g., tofacitinib, baricitinib, filgotinib, upadacitinib).
* Screening laboratory and other analyses show any prespecified abnormal hematologic results.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (379):
- United States (114):
  - East View Medical Research, LLC /ID# 216933, Mobile, Alabama
  - CB Flock Research Corporation /ID# 206094, Mobile, Alabama
  - Arizona Arthritis & Rheumatology Research, PLLC /ID# 211030, Sun City, Arizona
  - Digestive Disease Consultants, A Division of Arizona Digestive Health, P.C /ID# 211887, Tempe, Arizona
  - University of Arizona /ID# 208856, Tucson, Arizona
  - Citrus Valley Gastroenterology /ID# 205627, Covina, California
  - Care Access Research /ID# 217003, Huntington Beach, California
  - Moore UC San Diego Cancer Center /ID# 204919, La Jolla, California
  - United Medical Doctors /ID# 207867, Los Alamitos, California
  - TLC Clinical Research Inc /ID# 216831, Los Angeles, California
  - Gastrointestinal Biosciences Clinical Trials, LLC /ID# 205314, Los Angeles, California
  - Facey Medical Foundation /ID# 205301, Mission Hills, California
  - United Medical Doctors - Murrieta /ID# 205313, Murrieta, California
  - InSite Digestive Health Care - Oxnard /ID# 205628, Oxnard, California
  - Inland Empire Clinical Trials, LLC /ID# 216164, Rialto, California
  - San Diego Clinical Trials /ID# 212122, San Diego, California
  - Medical Assoc Research Grp /ID# 205626, San Diego, California
  - Delta Waves, Inc. /ID# 206170, Colorado Springs, Colorado
  - Western States Clinical Res /ID# 206091, Wheat Ridge, Colorado
  - Western Connecticut Medical Group /ID# 208290, Danbury, Connecticut
  - Gastroenterology Center of CT /ID# 208291, Hamden, Connecticut
  - Gastro Florida /ID# 206174, Clearwater, Florida
  - Universal Axon Clinical Research /ID# 213462, Doral, Florida
  - Palmetto Research, LLC /ID# 208293, Hialeah, Florida
  - Nature Coast Clinical Research - Inverness /ID# 206087, Inverness, Florida
  - Encore Borland-Groover Clinical Research /Id# 208128, Jacksonville, Florida
  - Cfagi Llc /Id# 207995, Maitland, Florida
  - University of Miami /ID# 215445, Miami, Florida
  - Coral Research Clinic /ID# 208292, Miami, Florida
  - Advanced Research Institute, Inc /ID# 206077, New Port Richey, Florida
  - Endoscopic Research, Inc. /ID# 207360, Orlando, Florida
  - Omega Research Consultants /ID# 206066, Orlando, Florida
  - Clinical Research Trials of Florida, Inc. /ID# 206068, Tampa, Florida
  - University of South Florida /ID# 214495, Tampa, Florida
  - AdventHealth Tampa /ID# 207363, Tampa, Florida
  - Gastroenterology Associates of Central Georgia, LLC /ID# 216940, Macon, Georgia
  - Infinite Clinical Trials /ID# 215343, Riverdale, Georgia
  - Atlanta Gastroenterology Spec /ID# 206173, Suwanee, Georgia
  - Next Innovative Clinical Research - Chicago /ID# 217324, Chicago, Illinois
  - The University of Chicago Medical Center /ID# 206172, Chicago, Illinois
  - Carle Foundation Hospital /ID# 207397, Effingham, Illinois
  - MediSphere Medical Research Center /ID# 206073, Evansville, Indiana
  - Indianapolis Gastroenterology /ID# 206381, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics /ID# 206167, Iowa City, Iowa
  - Cotton-O'Neil Clinical Res Ctr /ID# 206175, Topeka, Kansas
  - Tri-State Gastroenterology /ID# 206124, Crestview Hills, Kentucky
  - Houma Digestive Health Special /ID# 206176, Houma, Louisiana
  - Louisana Research Center, LLC /ID# 206064, Shreveport, Louisiana
  - Gastro Center of Maryland /ID# 206883, Columbia, Maryland
  - University of Michigan Health Systems /ID# 206918, Ann Arbor, Michigan
  - Huron Gastroenterology Assoc /ID# 205109, Ann Arbor, Michigan
  - Clin Res Inst of Michigan, LLC /ID# 207078, Chesterfield, Michigan
  - Revival Research Institute, LLC /ID# 207282, Southfield, Michigan
  - Center for Digestive Health /ID# 207080, Troy, Michigan
  - Mayo Clinic /ID# 205645, Rochester, Minnesota
  - University of Mississippi Medical Center /ID# 213116, Jackson, Mississippi
  - Southern Therapy and Advanced Research (STAR) LLC /ID# 206069, Jackson, Mississippi
  - Las Vegas Medical Research /ID# 206814, Las Vegas, Nevada
  - AGA Clinical Research Associates, LLC /ID# 206880, Egg Harbor, New Jersey
  - Atlantic Digestive Health Inst /ID# 208748, Morristown, New Jersey
  - Rutgers Robert Wood Johnson /ID# 207382, New Brunswick, New Jersey
  - University of New Mexico Department of Internal Medicine /ID# 214397, Albuquerque, New Mexico
  - NY Scientific /ID# 206080, Brooklyn, New York
  - NYU Langone Long Island Clinical Research Associates /ID# 206079, Lake Success, New York
  - DiGiovanna Institute for Medical Education & Research /ID# 206885, North Massapequa, New York
  - Premier Medical Group - GI Division /ID# 206097, Poughkeepsie, New York
  - Gastro Group of Rochester /ID# 206881, Rochester, New York
  - Richmond University Medical Center /ID# 213185, Staten Island, New York
  - Advantage Clinical Trials /ID# 206082, The Bronx, New York
  - Digestive Health Partners, P.A /ID# 206842, Asheville, North Carolina
  - Atrium Health Carolinas Medical Center /ID# 206085, Charlotte, North Carolina
  - Charlotte Gastroenterology and Hepatology, PLLC /ID# 206138, Charlotte, North Carolina
  - Wake Forest Baptist Medical Center /ID# 206067, Winston-Salem, North Carolina
  - Duplicate_Plains Clinical Research Center, LLC /ID# 205111, Fargo, North Dakota
  - University of Cincinnati /ID# 205633, Cincinnati, Ohio
  - The Ohio State University /ID# 205637, Columbus, Ohio
  - Optimed Research, Ltd. /ID# 205638, Columbus, Ohio
  - Hometown Urgent Care and Resea /ID# 205630, Dayton, Ohio
  - Dayton Gastroenterology, Inc. /ID# 205639, Englewood, Ohio
  - Great Lakes Gastroenterology Research LLC /ID# 205631, Mentor, Ohio
  - Hightower Clinical /ID# 216336, Oklahoma City, Oklahoma
  - Digestive Disease Specialists /ID# 206076, Oklahoma City, Oklahoma
  - Options Health Research, LLC /ID# 206707, Tulsa, Oklahoma
  - Healthcare Research Consultant /ID# 206706, Tulsa, Oklahoma
  - Guthrie Medical Group, PC /ID# 206078, Sayre, Pennsylvania
  - Pharmacorp Clinical Trials /ID# 206074, Charleston, South Carolina
  - Gastroenterology Associates, P.A. of Greenville /ID# 206098, Greenville, South Carolina
  - Gastro One /ID# 206178, Germantown, Tennessee
  - East Tennessee Research Institute /ID# 206169, Johnson City, Tennessee
  - Quality Medical Research /ID# 206088, Nashville, Tennessee
  - Vanderbilt University Medical Center /ID# 210405, Nashville, Tennessee
  - TX Clinical Research Institute /ID# 206718, Arlington, Texas
  - Inquest Clinical Research /ID# 206132, Baytown, Texas
  - Texas Digestive Disease Consultants /ID# 209805, Cedar Park, Texas
  - Texas Digestive Disease Consultants /ID# 209948, Cedar Park, Texas
  - Baylor Scott & White Center for Inflammatory Bowel Diseases /ID# 207484, Dallas, Texas
  - DHAT Research Institute /ID# 206716, Garland, Texas
  - Vilo Research Group Inc /ID# 212625, Houston, Texas
  - Baylor College of Medicine - Baylor Medical Center /ID# 206717, Houston, Texas
  - Centex Studies, Inc. - Houston /ID# 206168, Houston, Texas
  - GI Specialists of Houston /ID# 206090, Houston, Texas
  - Caprock Gastro Research /ID# 215115, Lubbock, Texas
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 206710, San Antonio, Texas
  - Southern Star Research Institute, LLC /ID# 205379, San Antonio, Texas
  - Baylor Scott & White Center for Diagnostic Medicine /ID# 206096, Temple, Texas
  - Duplicate_Tyler Research Institue /ID# 206075, Tyler, Texas
  - Gastro Health & Nutrition - Victoria /ID# 205378, Victoria, Texas
  - Advanced Research Institute /ID# 206133, Ogden, Utah
  - Ctr for Gastrointestinal Healt /ID# 208475, Franklin, Virginia
  - Washington Gastroenterology Associates /ID# 206177, Bellevue, Washington
  - Virginia Mason - Seattle Orthapedics /ID# 206070, Seattle, Washington
  - The Vancouver Clinic, INC. PS /ID# 204973, Vancouver, Washington
  - Wisconsin Center for Advanced Research, a division of GI Associates, LLC /ID# 206917, Milwaukee, Wisconsin
  - Froedtert Memorial Lutheran Hospital /ID# 206945, Milwaukee, Wisconsin
- Argentina (5):
  - Cardio Alem /ID# 211282, San Isidro, Buenos Aires
  - Mautalen Salud e Investigacion /ID# 206033, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Hospital Britanico de Buenos Aires /ID# 209497, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Gedyt /ID# 210017, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Hospital Privado Univesitario /ID# 206030, Córdoba
- Australia (6):
  - Macquarie University Hospital /ID# 211955, Macquarie University, New South Wales
  - Duplicate_Mater Misericordiae /ID# 212687, South Brisbane, Queensland
  - Griffith University /ID# 211956, Southport, Queensland
  - St Vincent's Hospital Melbourne /ID# 205758, Fitzroy, Victoria
  - Monash Medical Centre /ID# 206486, Melbourne, Victoria
  - Fiona Stanley Hospital /ID# 211642, Murdoch, Western Australia
- Austria (3):
  - Klinik Landstrasse /ID# 205764, Vienna, Vienna
  - Medical University of Vienna /ID# 205763, Vienna, Vienna
  - LKH Salzburg and Paracelsus /ID# 208788, Salzburg
- Belgium (2):
  - Universitair Ziekenhuis Leuven /ID# 205988, Leuven, Vlaams-Brabant
  - AZ Maria Middelares /ID# 210928, Ghent
- Bosnia and Herzegovina (5):
  - University Clinical Centre of the Republic of Srpska /ID# 208053, Banja Luka, Republika Srpska
  - University Clinical Centre of the Republic of Srpska /ID# 208055, Banja Luka, Republika Srpska
  - University Clinical Center Tuzla /ID# 208057, Tuzla, Tuzlanski
  - University Clinical Hospital Mostar /ID# 208054, Mostar
  - Clinical Center University of Sarajevo /ID# 208058, Sarajevo
- Brazil (6):
  - Hospital Nossa Senhora das Graças /ID# 206981, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 206985, Porto Alegre, Rio Grande do Sul
  - Upeclin Fmb - Unesp /Id# 206986, Botucatu, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto - USP /ID# 206504, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC /ID# 206984, Santo André, São Paulo
  - Kaiser Clinica e Hospital Dia /ID# 206982, São José do Rio Preto, São Paulo
- Canada (7):
  - University of Calgary - Cumming School of Medicine - Adult Cystic Fibrosis Clini /ID# 205755, Calgary, Alberta
  - Allen Whey Khye Lim Professional Corporation /ID# 211167, Edmonton, Alberta
  - Covenant Health /ID# 205500, Edmonton, Alberta
  - Percuro Clinical Research, Ltd /ID# 205501, Victoria, British Columbia
  - Duplicate_Toronto Digestive Disease Asso /ID# 205498, Vaughan, Ontario
  - Crchum /Id# 207387, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS /ID# 205499, Sherbrooke, Quebec
- Chile (5):
  - Research Group /ID# 208037, Santiago, Santiago Metropolitan
  - M y F Estudios Clínicos Ltda. /ID# 208035, Santiago, Santiago Metropolitan
  - Hospital Guillermo Grant Benavente de Concepción /ID# 212426, Concepción
  - CTR Estudios Clinicos /ID# 208036, Providencia
  - Hospital Clinico Universidad De Los Andes /ID# 207426, Santiago
- China (11):
  - Sun Yat-sen Memorial Hospital of Sun Yat-sen University /ID# 205267, Guangzhou, Guangdong
  - The Sixth Affiliated Hosp Sun /ID# 205268, Guangzhou, Guangdong
  - Affiliated Taihe Hospital of Hubei University of Medicine /ID# 216406, Shiyan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 205266, Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University /ID# 212186, Nanchang, Jiangxi
  - The First Hospital of Jilin University /ID# 210088, Changchun, Jilin
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 205333, Shanghai, Shanghai Municipality
  - The second Affiliated hospital of Zhejiang University school of Medicine /ID# 205271, Hangzhou, Zhejiang
  - West China Hospital, Sichuan University /ID# 205332, Chengdu
  - Duplicate_Tianjin Med Univ General Hosp /ID# 205246, Tianjin
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Techno /ID# 205265, Wuhan
- Colombia (3):
  - Corporacion Hospitalaria Juan Cuidad Sede Denominada Hospital Universitario Mayo /ID# 208886, Bogota DC, Cundinamarca
  - Instituto Medico de Alta Tecnologia Oncomédica S.A /ID# 208887, Montería, Departamento de Córdoba
  - Hospital Universitario San Vic /ID# 208888, Medellín
- Croatia (4):
  - Klinicka bolnica Dubrava Zagreb /ID# 208460, Zagreb, City of Zagreb
  - Poliklinika Solmed /ID# 211568, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Rijeka /ID# 208650, Rijeka, Primorje-Gorski Kotar County
  - Klinicki bolnicki centar Split /ID# 217027, Split
- Czechia (7):
  - Hepato-Gastroenterologie HK, s.r.o. /ID# 205672, Hradec Králové
  - CTCenter MaVe s.r.o. /ID# 205671, Olomouc
  - Artroscan s.r.o. /ID# 205668, Ostrava
  - Nemocnice Pardubickeho kraje, a.s. /ID# 213540, Pardubice
  - Nemocnice Milosrdnych sester sv. Karla Boromejskeho v Praze /ID# 216223, Prague
  - Axon Clinical, s.r.o. /ID# 205670, Prague
  - ISCARE a.s. /ID# 209240, Prague
- Estonia (4):
  - East Tallinn Central Hospital /ID# 207564, Tallinn, Harju
  - West Tallinn Central Hospital /ID# 207356, Tallinn
  - North Estonia Medical Centre /ID# 207357, Tallinn
  - Tartu University Hospital /ID# 212282, Tartu
- Finland (4):
  - Tampere University Hospital /ID# 206161, Tampere, Pirkanmaa
  - Keski-Suomen Sairaala Nova /ID# 206159, Jyväskylä
  - Laakarikeskus Ikioma /ID# 205814, Mikkeli
  - Tyks /Id# 205813, Turku
- France (2):
  - Chu de Nice-Hopital L'Archet Ii /Id# 209118, Nice, Alpes-Maritimes
  - Centre Hospitalier Lyon Sud /ID# 209121, Pierre-Bénite, Rhone
- Germany (8):
  - Universitatsklinikum Mannheim /ID# 206811, Mannheim, Baden-Wurttemberg
  - Duplicate_Universitaetsklinikum Tuebingen /ID# 206737, Tübingen, Baden-Wurttemberg
  - Gastroenterologische Gemeinschaftspraxis Herne /ID# 214576, Herne, North Rhine-Westphalia
  - Zentrum für Gastroenterologie Saar MVZ GmbH /ID# 215813, Saarbrücken, Saarland
  - Duplicate_Praxis am Bayrischen Platz /ID# 206733, Berlin
  - Agaplesion Markus Krankenhaus /ID# 206731, Frankfurt am Main
  - Duplicate_Univ Hosp Schleswig-Holstein /ID# 206791, Kiel
  - Medizinisches Versorgungszentrum Portal 10 /ID# 207137, Münster
- Greece (4):
  - General Hospital of Athens Laiko /ID# 208671, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 207061, Heraklion, Crete
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 206332, Athens
  - Duplicate_General Hospital of Thessaloniki Hippokrateio /ID# 208822, Thessaloniki
- Hungary (4):
  - Bekes Megyei Kozponti Korhaz /ID# 205885, Békéscsaba
  - Semmelweis Egyetem /ID# 205883, Budapest
  - Soproni Erzsebet Oktato Korhaz es Rehabilitacios Intezet /ID# 207992, Sopron
  - Mentahaz Maganorvosi Kozpont /ID# 205882, Székesfehérvár
- Ireland (2):
  - Beaumont Hospital /ID# 206509, Dublin
  - University Hospital Galway /ID# 218035, Galway
- Israel (2):
  - Rambam Health Care Campus /ID# 206362, Haifa
  - Shaare Zedek Medical Center /ID# 206365, Jerusalem
- Italy (7):
  - A.O.U. Policlinico S.Orsola-Malpighi /ID# 206351, Bologna, Emilia-Romagna
  - ASST Rhodense/Presidio Ospedaliero di Rho /ID# 216611, Rho, Milano
  - Istituto Clinico Humanitas /ID# 206346, Rozzano, Milano
  - Presidio Columbus-Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Un /ID# 206347, Rome, Roma
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 206354, Negrar, Verona
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 206349, Milan
  - A.O. Ospedali Riuniti Villa Sofia - Cervello /ID# 206350, Palermo
- Japan (62):
  - Nagoya University Hospital /ID# 206355, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 206058, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital /ID# 207625, Toyohashi, Aichi-ken
  - Ieda Hospital /ID# 207479, Toyota-shi, Aichi-ken
  - Hirosaki National Hospital /ID# 206387, Hirosaki-shi, Aomori
  - Tokatsu Tsujinaka Hospital /ID# 214963, Abiko-shi, Chiba
  - Tsujinaka Hospital Kashiwanoha /ID# 209573, Kashiwa-shi, Chiba
  - Toho University Medical Center Sakura Hospital /ID# 207705, Sakura-shi, Chiba
  - Juntendo University Urayasu Hospital /ID# 208784, Urayasu-shi, Chiba
  - Fukui Prefectural Hospital /ID# 210449, Fukui-shi, Fukui
  - Fukuoka University Chikushi Hospital /ID# 214405, Chikushino-shi, Fukuoka
  - Saiseikai Fukuoka Genaral Hospital /ID# 209482, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 206385, Kurume-shi, Fukuoka
  - Ogaki Municipal Hospital /ID# 208227, Ogaki-shi, Gifu
  - NHO Fukuyama Medical Center /ID# 206295, Fukuyama-shi, Hiroshima
  - Hiroshima University Hospital /ID# 206464, Hiroshima, Hiroshima
  - Asahikawa Medical University Hospital /ID# 206404, Midorigaokahiga-shi, Hokkaido
  - Obihiro kosei Hospital /ID# 210424, Obihiro-shi, Hokkaido
  - Sapporo Tokushukai Hospital /ID# 209448, Sapporo, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 206059, Sapporo, Hokkaido
  - Sapporo Medical University Hospital /ID# 206314, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital /ID# 208494, Sapporo, Hokkaido
  - Aoyama Clinic /ID# 206452, Kobe, Hyōgo
  - Hyogo College of Medicine Hospital /ID# 206455, Nishinomiya-shi, Hyōgo
  - Kanazawa University Hospital /ID# 206316, Kanazawa, Ishikawa-ken
  - Iwate Medical University Uchimaru Medical Center /ID# 207051, Morioka, Iwate
  - Idzuro Imamura Hospital /ID# 207639, Kagoshima, Kagoshima-ken
  - Sameshima Hospital /ID# 207935, Kagoshima, Kagoshima-ken
  - St. Marianna University School of Medicine Hospital /ID# 209451, Kawasaki-shi, Kanagawa
  - Showa University Fujigaoka Hospital /ID# 208224, Yokohama, Kanagawa
  - Kyoto University Hospital /ID# 211809, Kyoto, Kyoto
  - Mie University Hospital /ID# 206803, Tsu, Mie-ken
  - Yokkaichi Hazu Medical Center /ID# 214348, Yokkaichi-shi, Mie-ken
  - National Hospital Organization Sendai Medical Center /ID# 209528, Sendai, Miyagi
  - NHO Nagasaki Medical Center /ID# 210822, Omura-shi, Nagasaki
  - Kenseikai Dongo Hospital /ID# 208101, Yamatotakada-shi, Nara
  - Saiseikai Niigata Hospital /ID# 209921, Niigata, Niigata
  - Niigata University Medical & Dental Hospital /ID# 218049, Niigata, Niigata
  - Ishida Clinic of IBD and Gastroenterology /ID# 210119, Ōita, Oita Prefecture
  - Chikuba Hospital for Proctological and Gastrointestinal Diseases /ID# 206646, Kurashiki-shi, Okayama-ken
  - Okayama University Hospital /ID# 217925, Okayama, Okayama-ken
  - Kinshukai Infusion Clinic /ID# 207865, Osaka, Osaka
  - Kitano Hospital /ID# 210397, Osaka, Osaka
  - Japanese Red Cross Osaka Hospital /ID# 209478, Osaka, Osaka
  - Osaka City University Hospital /ID# 206457, Osaka, Osaka
  - Toyonaka Municipal Hospital /ID# 217082, Toyonaka-shi, Osaka
  - Saga University Hospital /ID# 209270, Saga, Saga-ken
  - Saitama Medical Center /ID# 206393, Kawagoe-shi, Saitama
  - Tokitokai Tokito clinic /ID# 206313, Saitama-shi, Saitama
  - National Hospital Organization Higashi-Ohmi General Medical Center /ID# 210710, Higashi-ohmi-shi, Shiga
  - Shimane University School of Medicine /ID# 208905, Izumo-shi, Shimane
  - Hamamatsu University Hospital /ID# 206459, Hamamatsu, Shizuoka
  - NHO Shizuoka Medical Center /ID# 208785, Sunto-gun, Shizuoka
  - Tokyo Medical And Dental University, Medical Hospital /ID# 206453, Bunkyo-ku, Tokyo
  - St.Luke's International Hospital /ID# 208076, Chuo-ku, Tokyo
  - Tokai University Hachioji Hospital /ID# 208903, Hachioji-shi, Tokyo
  - Teikyo University Hospital /ID# 209866, Itabashi-ku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine /ID# 209532, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 206460, Shinjuku-ku, Tokyo
  - Yamagata University Hospital /ID# 206465, Yamagata, Yamagata
  - Tokuyama Central Hospital /ID# 216994, Shunan-shi, Yamaguchi
  - Shoyukai Fujita Gastroenterological Hospital /ID# 216493, Takatsuki-shi
- Latvia (2):
  - Riga East Clinical Univ Hosp /ID# 206828, Riga
  - P. Stradins Clinical Univ Hosp /ID# 206827, Riga
- Lithuania (4):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 209052, Kaunas
  - Klaipeda Seamens Hospital /ID# 208791, Klaipėda
  - Klaipeda University Hospital /ID# 208790, Klaipėda
  - Vilnius University Hospital /ID# 209051, Vilnius
- Malaysia (2):
  - Universiti Kebangsaan Malaysia (UKM) Medical Centre /ID# 207662, Kuala Lumpur, Selangor
  - Duplicate_Uni Malaya MC /ID# 208936, Kuala Lumpur
- Mexico (3):
  - Morales Vargas Centro de Investigacion S.C. /ID# 211326, León, Guanajuato
  - Clinica de Investigacion en Reumatologia y Obesidad S.C. /ID# 208068, Guadalajara, Jalisco
  - Centro Regiomontano de Estudios Clínicos ROMA S.C /ID# 208067, Monterrey, Nuevo León
- Erasmus Medisch Centrum /ID# 205280, Rotterdam, Netherlands
- Norway (2):
  - Akershus Universitetssykehus_MAIN /ID# 205293, Lorenskog, Akershus
  - Universitetssykehuset Nord-Norge /ID# 205691, Tromsø, Troms
- Poland (6):
  - Gastromed /Id# 216108, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Zdrowia MDM /ID# 205874, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Reuma Park w Warszawie /ID# 212913, Warsaw, Masovian Voivodeship
  - NZOZ Vivamed /ID# 216697, Warsaw, Masovian Voivodeship
  - Instytut Pomnik - Centrum Zdrowia Dziecka /ID# 215070, Warsaw, Masovian Voivodeship
  - Endoskopia Sp. z o.o. /ID# 212964, Sopot, Pomeranian Voivodeship
- Portugal (8):
  - Hospital da Senhora da Oliveira Guimaraes, EPE /ID# 205554, Guimarães, Braga District
  - Centro Hospitalar de Entre Douro e Vouga /ID# 205563, Santa Maria DA Feira, Porto District
  - Unidade Local de Saúde do Alto Minho, EPE - Hospital Conde de Bertiandos /ID# 205556, Ponte de Lima, Viana do Castelo District
  - Hospital Garcia de Orta, EPE /ID# 206143, Almada
  - CCA Braga - Hospital de Braga /ID# 206144, Braga
  - Hospital Santo Antonio dos Cap /ID# 206145, Lisbon
  - Centro Hospitalar Universitário de Lisboa Norte, EPE - Hospital de Santa Maria /ID# 206117, Lisbon
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 206142, Porto
- School of Medicine University of Puerto Rico-Medical Science Campus /ID# 209626, San Juan, Puerto Rico
- Russia (10):
  - Immanuel Kant Baltic Federal University /ID# 208264, Kaliningrad, Kaliningrad Oblast
  - NW State Medical Univ na Mechn /ID# 208258, Saint Petersburg, Leningradskaya Oblast'
  - Perm Clinical Center of the Federal Medical and Biological Agency /ID# 211653, Perm, Permskiy Kray
  - Medical Company Hepatolog /ID# 208261, Samara, Samara Oblast
  - Professor Pasechnikov Gastroenterology and Pankreatology clinic /ID# 211652, Stavropol, Stavropol Kray
  - Kazan State Medical University /ID# 208256, Kazan', Tatarstan, Respublika
  - Olla-Med Clinic /ID# 215335, Moscow
  - Republican hospital named after V.A. Baranov /ID# 206507, Petrozavodsk
  - Euromedservice /ID# 208265, Pushkin
  - LLC Novaya Clinica /ID# 208260, Pyatigorsk
- Serbia (8):
  - Clinical Hosp Center Zvezdara /ID# 205258, Belgrade, Beograd
  - Military Medical Academy /ID# 205257, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 205256, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 206413, Belgrade, Beograd
  - University Clinical Center of Nis /ID# 206411, Niš, Nisavski Okrug
  - University Clinical Center Kragujevac /ID# 206410, Kragujevac, Sumadijski Okrug
  - Clinical Center Vojvodina /ID# 205259, Novi Sad, Vojvodina
  - General Hospital Leskovac /ID# 217881, Leskovac
- Singapore (3):
  - National University Hospital /ID# 209099, Singapore
  - Gleneagles Medical Centre /ID# 206954, Singapore
  - Tan Tock Seng Hospital /ID# 207663, Singapore
- Slovakia (5):
  - Medak s.r.o. /ID# 205191, Bratislava, Bratislava Region
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 205147, Banská Bystrica
  - B+B MED, s.r.o. /ID# 205213, Košice
  - Fakultna nemocnica s poliklini /ID# 211372, Nové Zámky
  - GASTRO I., s.r.o. /ID# 205148, Prešov
- South Africa (8):
  - MD Search /ID# 208084, Boksburg North, Gauteng
  - Clinresco Centers /ID# 208083, Johannesburg, Gauteng
  - Lenasia Clinical Trial Centre /ID# 214359, Johannesburg, Gauteng
  - Wits Clinical Research , Wits Health Consortium (PTY) Ltd /ID# 208082, Johannesburg, Gauteng
  - Wits Clinical Research Site /ID# 208949, Johannesburg, Gauteng
  - Kingsbury Hospital /ID# 205281, Cape Town, Western Cape
  - Private Practice Dr MN Rajabally /ID# 205273, Cape Town, Western Cape
  - Mediclinic Milnerton /ID# 207979, CAPE TOWN Milnerton, Western Cape
- South Korea (6):
  - Kangbuk Samsung Hospital /ID# 206960, Seoul, Seoul Teugbyeolsi
  - Dong-A University Hospital /ID# 206955, Busan
  - Pusan National University Hospital /ID# 206956, Busan
  - Yeungnam University Medical Center /ID# 206959, Daegu
  - Duplicate_CHA Bundang Medical Center /ID# 207432, Seongnam-si, Gyeonggi-do
  - Yonsei University Health System, Severance hospital /ID# 206958, Seoul
- Spain (10):
  - Hospital Clínico Universitario de Santiago-CHUS /ID# 204411, Santiago de Compostela, A Coruna
  - Hospital Unversitario Marques de Valdecilla /ID# 216622, Santander, Cantabria
  - Hospital Universitario Dr. Negrin /ID# 206905, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario A Coruna - CHUAC /ID# 206907, A Coruña
  - Hospital Clinic de Barcelona /ID# 206906, Barcelona
  - Hospital Universitario Reina Sofia /ID# 204412, Córdoba
  - Hospital Universitario Ramon y Cajal /ID# 204410, Madrid
  - Hospital Universitario La Paz /ID# 214540, Madrid
  - Hospital Clinico Universitario de Salamanca /ID# 205013, Salamanca
  - Hospital Universitario y Politecnico La Fe /ID# 206904, Valencia
- Switzerland (4):
  - Kantonsspital St. Gallen /ID# 211310, Sankt Gallen, Canton of St. Gallen
  - Universitaetsspital Basel /ID# 211381, Basel
  - Inselspital, Universitaetsklinik /ID# 211312, Bern
  - Universitaetsspital Zuerich /ID# 211308, Zurich
- Taiwan (4):
  - China Medical University Hosp /ID# 207845, Taichung, Taichung
  - National Taiwan University Hospital /ID# 207847, Taipei City, Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 207848, Kaohsiung City
  - Taipei Veterans General Hosp /ID# 207849, Taipei
- Turkey (Türkiye) (5):
  - Erciyes University Medical Fac /ID# 207506, Melikgazi, Kayseri
  - Gazi University Med. Faculty /ID# 208040, Ankara GAZI
  - Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty /ID# 207507, Istanbul
  - Umraniye Training and Res Hosp /ID# 208206, Istanbul
  - Mersin University Medical /ID# 208039, Mersin
- Ukraine (5):
  - Communal Non-Commercial Enterprize of Kharkiv Regional Council Regional Clinical /ID# 206939, Kharkiv, Kharkivs’ka Oblast’
  - Kyiv Regional Hospital /ID# 217373, Kyiv, Kyivska Oblast
  - PE PMC Acinus, Medical and Diagnostic Center /ID# 217218, Kropyvnytskyi
  - Medical centre of CONSILIUM MEDICAL LLC /ID# 217447, Kyiv
  - Vinnytsia Regional Clinical Hospital n.a. M.I.Pyrogov /ID# 216300, Vinnytsia
- United Kingdom (5):
  - Basingstoke & North Hampshire /ID# 207985, Basingstoke
  - Queen Elizabeth University Hos /ID# 205154, Glasgow
  - Huddersfield Royal Infirmary /ID# 217660, Huddersfield
  - St. George's Healthcare NHS /ID# 208375, London
  - Barts and the London NHS Trust /ID# 205153, Whitechapel

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Vermeire S, Colombel JF, Danese S, Panaccione R, Peyrin-Biroulet L, Beck K, Chaparro M, Gisbert JP, Dubcenco E, Klaff J, Naling G, Ford S, Remple V, Joshi N, Suravaram S, Duncan B, Wang Y, Wick-Urban B, Loftus EV. Benefit-risk profile of upadacitinib: exploratory post hoc analysis of phase 2b/3 studies in patients with moderately to severely active ulcerative colitis or Crohn's disease. J Crohns Colitis. 2026 Jan 9;20(1):jjaf198. doi: 10.1093/ecco-jcc/jjaf198. PMID 41264726
- [Derived] Panes J, Dubinsky MC, Ishiguro Y, Shukla N, Dubcenco E, Remple V, Sharma D, Panaccione R. Achievement of long-term treatment goals in upadacitinib-treated patients with moderately to severely active ulcerative colitis: a post hoc analysis of phase 3 trial data. J Crohns Colitis. 2025 Jul 3;19(7):jjaf095. doi: 10.1093/ecco-jcc/jjaf095. PMID 40488552
- [Derived] Panaccione R, Danese S, Zhou W, Klaff J, Ilo D, Yao X, Levy G, Higgins PDR, Loftus EV Jr, Chen S, Gonzalez YS, Leonard C, Hebuterne X, Lindsay JO, Cao Q, Nakase H, Colombel JF, Vermeire S. Efficacy and safety of upadacitinib for 16-week extended induction and 52-week maintenance therapy in patients with moderately to severely active ulcerative colitis. Aliment Pharmacol Ther. 2024 Feb;59(3):393-408. doi: 10.1111/apt.17816. Epub 2023 Nov 27. PMID 38010661
- [Derived] Raine T, Ishiguro Y, Rubin DT, Finney-Hayward T, Vladea R, Liu J, Phillips C, Cheng E, Targownik L, Loftus EV Jr. Impact of Baseline Corticosteroid Use on the Efficacy and Safety of Upadacitinib in Patients with Ulcerative Colitis: A Post Hoc Analysis of the Phase 3 Clinical Trial Programme. J Crohns Colitis. 2024 May 31;18(5):695-707. doi: 10.1093/ecco-jcc/jjad190. PMID 37942921
- [Derived] Danese S, Tran J, D'Haens G, Rubin DT, Aoyama N, Zhou W, Ilo D, Yao X, Sanchez Gonzalez Y, Panaccione R. Upadacitinib Induction and Maintenance Therapy Improves Abdominal Pain, Bowel Urgency, and Fatigue in Patients With Ulcerative Colitis: A Post Hoc Analysis of Phase 3 Data. Inflamm Bowel Dis. 2023 Nov 2;29(11):1723-1729. doi: 10.1093/ibd/izad016. PMID 36790041
- [Derived] Panes J, Loftus EV, Higgins PDR, Lindsay JO, Zhou W, Yao X, Ilo D, Phillips C, Tran J, Sanchez Gonzalez Y, Vermeire S. Induction and Maintenance Treatment With Upadacitinib Improves Health-Related Quality of Life in Patients With Moderately to Severely Active Ulcerative Colitis: Phase 3 Study Results. Inflamm Bowel Dis. 2023 Sep 1;29(9):1421-1430. doi: 10.1093/ibd/izac260. PMID 36645051
- [Derived] Ponce-Bobadilla AV, Stodtmann S, Eckert D, Zhou W, Liu W, Mohamed MF. Upadacitinib Population Pharmacokinetics and Exposure-Response Relationships in Ulcerative Colitis Patients. Clin Pharmacokinet. 2023 Jan;62(1):101-112. doi: 10.1007/s40262-022-01191-6. Epub 2022 Dec 26. PMID 36571701
- [Derived] Loftus EV Jr, Colombel JF, Takeuchi K, Gao X, Panaccione R, Danese S, Dubinsky M, Schreiber S, Ilo D, Finney-Hayward T, Zhou W, Phillips C, Gonzalez YS, Shu L, Yao X, Zhou Q, Vermeire S. Upadacitinib Therapy Reduces Ulcerative Colitis Symptoms as Early as Day 1 of Induction Treatment. Clin Gastroenterol Hepatol. 2023 Aug;21(9):2347-2358.e6. doi: 10.1016/j.cgh.2022.11.029. Epub 2022 Dec 1. PMID 36464141
- [Derived] Danese S, Vermeire S, Zhou W, Pangan AL, Siffledeen J, Greenbloom S, Hebuterne X, D'Haens G, Nakase H, Panes J, Higgins PDR, Juillerat P, Lindsay JO, Loftus EV Jr, Sandborn WJ, Reinisch W, Chen MH, Sanchez Gonzalez Y, Huang B, Xie W, Liu J, Weinreich MA, Panaccione R. Upadacitinib as induction and maintenance therapy for moderately to severely active ulcerative colitis: results from three phase 3, multicentre, double-blind, randomised trials. Lancet. 2022 Jun 4;399(10341):2113-2128. doi: 10.1016/S0140-6736(22)00581-5. Epub 2022 May 26. PMID 35644166
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included a Screening Period of up to 5 weeks, Part 1, and Part 2. Part 1 was a randomized, double-blind, placebo-controlled 8-week induction period. Part 2 was an open-label, 8-week extended treatment period for participants who were clinical non-responders in Part 1.
  Participants with moderately to severely active ulcerative colitis (UC) were randomized at 204 sites in 41 countries.
Pre-assignment Details: In Part 1 participants were randomized in a 2:1 ratio to upadacitinib or placebo. Randomization was stratified by biologic-inadequate responder (Bio-IR) status (bio-IR vs non-bio-IR), corticosteroid use (yes or no), and Adapted Mayo score (≤ 7 or > 7) at Baseline. Within bio-IR, randomization was further stratified by number of prior biologic treatments (≤ 1 or > 1). Within non-bio-IR, randomization was further stratified by previous biologic use (yes or no).
Groups:
- Part 1: Upadacitinib 45 mg: Participants received 45 mg upadacitinib once daily (QD) for 8 weeks.
- Part 1: Placebo: Participants received placebo matching to upadacitinib once daily for 8 weeks.
- Part 2: Upadacitinib 45 mg / Upadacitinib 45 mg: Participants initially assigned to upadacitinib who did not achieve clinical response per Adapted Mayo score at Week 8 in Part 1 received upadacitinib 45 mg once daily for 8 additional weeks in the open-label extension period.
- Part 2: Placebo / Upadacitinib 45 mg: Participants initially assigned to placebo who did not achieve clinical response per Adapted Mayo score at Week 8 in Part 1 received upadacitinib 45 mg once daily for 8 weeks in the open-label extension period.
Period: Part 1: Placebo-controlled Period
Arm/Group | Part 1: Upadacitinib 45 mg | Part 1: Placebo | Part 2: Upadacitinib 45 mg / Upadacitinib 45 mg | Part 2: Placebo / Upadacitinib 45 mg
Started | 345 | 177 | 0 | 0
Received Treatment | 344 | 177 | 0 | 0
Completed | 334 | 164 | 0 | 0
Not Completed | 11 | 13 | 0 | 0
Not completed — Adverse Event | 5 | 6 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 0 | 0
Not completed — Other | 0 | 3 | 0 | 0
Period: Part 2: Open-label Extension
Arm/Group | Part 1: Upadacitinib 45 mg | Part 1: Placebo | Part 2: Upadacitinib 45 mg / Upadacitinib 45 mg | Part 2: Placebo / Upadacitinib 45 mg
Started (Part 2 was an extended treatment period for participants who did not achieve clinical response per Adapted Mayo score at Week 8 in Part 1.) | 0 | 0 | 68 | 116
Completed | 0 | 0 | 65 | 111
Not Completed | 0 | 0 | 3 | 5
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Other | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Upadacitinib 45 mg: Participants received 45 mg upadacitinib once daily (QD) for 8 weeks.
- Placebo: Participants received placebo matching to upadacitinib once daily for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Upadacitinib 45 mg | Placebo | Total
Number analyzed (Participants) | 345 | 177 | 522
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (14.73) | 42.2 (14.44) | 42.2 (14.62)
Age, Customized [Count of Participants; unit: Participants]
  < 18 years | 6 | 3 | 9
  ≥ 18 years to < 40 years | 160 | 81 | 241
  ≥ 40 years to < 65 years | 146 | 79 | 225
  ≥ 65 years | 33 | 14 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 67 | 196
  Male | 216 | 110 | 326
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 16 | 42
  Not Hispanic or Latino | 319 | 161 | 480
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 238 | 127 | 365
  Black or African American | 11 | 6 | 17
  Asian | 94 | 41 | 135
  American Indian or Alaska Native | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Multiple | 2 | 1 | 3
Biologic-inadequate Responder (Bio-IR) Status [Count of Participants; unit: Participants] — Biologic-inadequate responders (Bio-IR) are defined as participants who had inadequate response, loss of response, or intolerance to biologic therapy.
  Non-biologic-inadequate responders (non-bio-IR) are defined as participants who had inadequate response, loss of response, or intolerance to conventional therapy but had not failed biologic therapy.
  Participants
    Bio-IR | 175 | 91 | 266
    Non-Bio-IR | 170 | 86 | 256
Baseline Corticosteroid Use [Count of Participants; unit: Participants]
  Yes | 123 | 75 | 198
  No | 222 | 102 | 324
Adapted Mayo Score Strata [Count of Participants; unit: Participants] — The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
  The overall Adapted Mayo Score ranges from 0 to 9 where higher scores represent more severe disease.
  Participants
    ≤ 7 | 205 | 104 | 309
    > 7 | 138 | 73 | 211
    Missing | 2 | 0 | 2
Bio-IR: Number of Prior Biologic Treatments [Count of Participants; unit: Participants] — Population: Biologic-inadequate responders
  Participants
    number analyzed (Participants) | 175 | 91 | 266
    ≤ 1 prior biologic | 58 | 33 | 91
    > 1 prior biologic | 117 | 58 | 175
Non-Bio-IR: Prior Exposure to Biologic Therapy [Count of Participants; unit: Participants] — Population: Non-biologic-inadequate responders
  Participants
    number analyzed (Participants) | 170 | 86 | 256
    Yes | 1 | 5 | 6
    No | 169 | 81 | 250
Disease Duration [Mean (Standard Deviation); unit: years] | 7.273 (6.4459) | 7.584 (7.6701) | 7.379 (6.8804)
Adapted Mayo Score [Mean (Standard Deviation); unit: units on a scale] — The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration). The overall score ranges from 0 to 9 where higher scores represent more severe disease. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 343 | 177 | 520
    (all) | 7.00 (1.216) | 7.05 (1.236) | 7.02 (1.222)
Average Stool Frequency Subscore [Mean (Standard Deviation); unit: units on a scale] — Participants recorded stool frequency using an electronic subject diary on a daily basis. The stool frequency subscore (SFS) ranges from 0 to 3 according to the following scale:
  Score 0: Normal number of stools
  Score 1: 1 to 2 stools more than normal
  Score 2: 3 to 4 stools more than normal
  Score 3: 5 or more stools more than normal Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 343 | 177 | 520
    (all) | 2.55 (0.626) | 2.64 (0.551) | 2.58 (0.603)
Average Rectal Bleeding Subscore [Mean (Standard Deviation); unit: units on a scale] — Participants recorded rectal bleeding in an electronic subject diary on a daily basis. The rectal bleeding subscore ranges from 0 to 3 according to the following scale:
  Score 0: No blood seen
  Score 1: Streaks of blood with stool less than half the time
  Score 2: Obvious blood with stool most of the time
  Score 3: Blood alone passed Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 343 | 177 | 520
    (all) | 1.77 (0.966) | 1.71 (1.049) | 1.75 (0.995)
Average Endoscopy Subscore [Mean (Standard Deviation); unit: units on a scale] — Findings on endoscopy were scored according to the following:
  Score 0: Normal or inactive disease
  Score 1: Mild disease (erythema, decreased vascular pattern)
  Score 2: Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions)
  Score 3: Severe disease (spontaneous bleeding, ulceration) Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 344 | 177 | 521
    (all) | 2.7 (0.47) | 2.7 (0.46) | 2.7 (0.46)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Remission Per Adapted Mayo Score at Week 8
Description: The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
  The overall Adapted Mayo score ranges from 0 to 9 where higher scores represent more severe disease.
  Clinical remission is defined as an Adapted Mayo score ≤ 2, with SFS ≤ 1 and not higher than Baseline, RBS of 0, and endoscopic subscore ≤ 1.
Time Frame: Week 8
Population: The Part 1 intent-to-treat population (ITT1) includes randomized participants who received at least 1 dose of study drug in Part 1. The ITT1 population excludes 6 participants from 1 site with non-compliance. Non-responder imputation incorporating multiple imputation to handle missing data due to Coronavirus Disease - 2019 (COVID-19) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Upadacitinib 45 mg: Participants received 45 mg upadacitinib once daily for 8 weeks.
Arm/Group | Upadacitinib 45 mg | Placebo
Number analyzed (Participants) | 341 | 174
percentage of participants | 33.5 [28.5 to 38.5] | 4.1 [1.1 to 7.1]
Statistical Analysis 1: Comparison: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The primary and ranked secondary efficacy endpoints were tested with multiplicity adjustment using a fixed-sequence multiple testing procedure to ensure a strong control of family-wise type I error rate at significance level alpha = 0.05 (2-sided); Adjusted for Baseline corticosteroid use (yes or no), Baseline Adapted Mayo score (≤ 7 or > 7), and bio-IR status (bio-IR or non-bio-IR); Adjusted Response Rate Difference = 29.0, 95% CI 2-sided [23.2 to 34.7] — Difference = Upadacitinib 45 mg - Placebo

2. Secondary Outcome: Percentage of Participants With Endoscopic Improvement at Week 8
Description: Endoscopic improvement is defined as an endoscopic subscore of 0 or 1. Endoscopies were assessed by a blinded central reader and scored according to the following scale: 0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern); 2 = Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration).
Time Frame: Week 8
Population: ITT1 population; non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Upadacitinib 45 mg | Placebo
Number analyzed (Participants) | 341 | 174
percentage of participants | 44.0 [38.8 to 49.3] | 8.3 [4.1 to 12.5]
Statistical Analysis 1: Comparison: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Response Rate Difference = 35.1, 95% CI 2-sided [28.6 to 41.6] — Difference = Upadacitinib 45 mg - Placebo

3. Secondary Outcome: Percentage of Participants With Endoscopic Remission at Week 8
Description: Endoscopic remission is defined as an endoscopic subscore of 0. Endoscopies were assessed by a blinded central reader and scored according to the following scale: 0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern); 2 = Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration).
Time Frame: Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Upadacitinib 45 mg | Placebo
Number analyzed (Participants) | 341 | 174
percentage of participants | 18.2 [14.1 to 22.3] | 1.7 [0.0 to 3.7]
Statistical Analysis 1: Comparison: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Response Rate Difference = 15.9, 95% CI 2-sided [11.4 to 20.3] — Difference = Upadacitinib 45 mg - Placebo

4. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response Per Adapted Mayo Score at Week 8
Description: The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease with spontaneous bleeding, ulceration).
  The overall Adapted Mayo score ranges from 0 to 9 with higher scores representing more severe disease.
  Clinical response per the Adapted Mayo Score is defined as a decrease in Adapted Mayo score ≥ 2 points and ≥ 30% from Baseline, plus a decrease in RBS ≥ 1 or an absolute RBS ≤ 1.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Upadacitinib 45 mg | Placebo
Number analyzed (Participants) | 341 | 174
percentage of participants | 74.5 [69.9 to 79.1] | 25.4 [18.9 to 31.8]
Statistical Analysis 1: Comparison: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Response Rate Difference = 49.4, 95% CI 2-sided [41.7 to 57.1] — Difference = Upadacitinib 45 mg - Placebo

5. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response Per Partial Adapted Mayo Score at Week 2
Description: The Partial Adapted Mayo Score is a composite score of UC disease activity based on the following 2 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  The overall Partial Adapted Mayo score ranges from 0 to 6 with higher scores representing more severe disease.
  Clinical response per Partial Adapted Mayo Score is defined as a decrease in Partial Adapted Mayo score ≥ 1 point and ≥ 30% from Baseline, plus a decrease in RBS ≥ 1 or an absolute RBS ≤ 1.
Time Frame: Week 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Upadacitinib 45 mg | Placebo
Number analyzed (Participants) | 341 | 174
percentage of participants | 63.3 [58.2 to 68.5] | 25.9 [19.4 to 32.4]
Statistical Analysis 1: Comparison: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Response Rate Difference = 37.0, 95% CI 2-sided [28.8 to 45.1] — Difference = Upadacitinib 45 mg - Placebo

6. Secondary Outcome: Percentage Of Participants Who Achieved Histologic-Endoscopic Mucosal Improvement at Week 8
Description: Histologic endoscopic mucosal improvement is defined as an endoscopic subscore of 0 or 1 and a Geboes score ≤ 3.1.
  The endoscopic subscore ranges from 0 (normal or inactive disease) to 3 (severe disease with spontaneous bleeding, ulceration).
  The Geboes histologic index includes seven histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades, each with 3-5 subgrades: Grade 0, structural change only; Grade 1, chronic inflammation; Grade 2, lamina propria neutrophils and eosinophils; Grade 3, neutrophils in epithelium; Grade 4, crypt destruction; and Grade 5, erosions or ulceration.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Upadacitinib 45 mg | Placebo
Number analyzed (Participants) | 341 | 174
percentage of participants | 36.7 [31.6 to 41.8] | 5.9 [2.3 to 9.4]
Statistical Analysis 1: Comparison: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Response Rate Difference = 30.1, 95% CI 2-sided [24.1 to 36.2] — Difference = Upadacitinib 45 mg - placebo

7. Secondary Outcome: Percentage of Participants Who Reported No Bowel Urgency at Week 8
Description: Bowel urgency was assessed by participants in a subject diary completed once a day.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Upadacitinib 45 mg | Placebo
Number analyzed (Participants) | 341 | 174
percentage of participants | 53.7 [48.4 to 59.0] | 25.9 [19.4 to 32.4]
Statistical Analysis 1: Comparison: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted for Baseline corticosteroid use (yes or no), Baseline Adapted Mayo score (<= 7 or > 7), and bio-IR status (bio-IR or non-bio-IR); Adjusted Response Rate Difference = 27.1, 95% CI 2-sided [19.0 to 35.3] — Difference = Upadacitinib 45 mg - Placebo

8. Secondary Outcome: Percentage of Participants Who Reported No Abdominal Pain at Week 8
Description: Abdominal pain was assessed by participants in a subject diary completed once a day.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Upadacitinib 45 mg | Placebo
Number analyzed (Participants) | 341 | 174
percentage of participants | 53.7 [48.4 to 59.0] | 24.1 [17.8 to 30.5]
Statistical Analysis 1: Comparison: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Response Rate Difference = 29.1, 95% CI 2-sided [20.9 to 37.4] — Difference = Upadacitinib 45 mg - Placebo

9. Secondary Outcome: Percentage of Participants Who Achieved Histologic Improvement at Week 8
Description: Histologic improvement is defined as a decrease from Baseline in Geboes score. The Geboes histologic index includes seven histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades, each with 3-5 subgrades: Grade 0, structural change only; Grade 1, chronic inflammation; Grade 2, lamina propria neutrophils and eosinophils; Grade 3, neutrophils in epithelium; Grade 4, crypt destruction; and Grade 5, erosions or ulceration.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Upadacitinib 45 mg | Placebo
Number analyzed (Participants) | 341 | 174
percentage of participants | 62.2 [57.0 to 67.3] | 24.5 [18.0 to 30.9]
Statistical Analysis 1: Comparison: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Response Rate Difference = 37.9, 95% CI 2-sided [29.8 to 46.1] — Difference = Upadacitinib 45 mg - Placebo

10. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Week 8
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) is used to assess health-related quality of life (HRQoL) in patients with ulcerative colitis. It consists of 32 questions evaluating bowel and systemic symptoms, as well as emotional and social functions. Each question is answered on a scale from 1 (worst) to 7 (best). The total score ranges from 32 to 224 with higher scores indicating better health-related quality of life. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Week 0) to Week 8
Population: ITT1 population with available data; a mixed effect model repeat measurement (MMRM) analysis with data from observed cases up to Week 8 was used except for measurements at or after the occurrence of UC-related corticosteroids intercurrent event were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Upadacitinib 45 mg | Placebo
Number analyzed (Participants) | 315 | 156
units on a scale | 52.2 [48.57 to 55.92] | 21.1 [15.98 to 26.17]
Statistical Analysis 1: Comparison: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed-effect model repeated measurement — [p-value comment as in outcome 1, analysis 1]; MMRM with Baseline, treatment, visit, treatment-by-visit interaction, and strata (Baseline Adapted Mayo score, corticosteroid use, and bio-IR status); Least Squares (LS) Mean Difference = 31.2, 95% CI 2-sided [24.98 to 37.36], Standard Error of Mean 3.15 — Difference = Upadacitinib 45 mg - Placebo

11. Secondary Outcome: Percentage of Participants Who Achieved Mucosal Healing at Week 8
Description: Mucosal healing is defined as an endoscopic score of 0 and Geboes score < 2.0. The endoscopic subscore ranges from 0 (normal or inactive disease) to 3 (severe disease with spontaneous bleeding, ulceration).
  The Geboes histologic index includes seven histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades, each with 3-5 subgrades: Grade 0, structural change only; Grade 1, chronic inflammation; Grade 2, lamina propria neutrophils and eosinophils; Grade 3, neutrophils in epithelium; Grade 4, crypt destruction; and Grade 5, erosions or ulceration.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Upadacitinib 45 mg | Placebo
Number analyzed (Participants) | 341 | 174
percentage of participants | 13.5 [9.9 to 17.1] | 1.7 [0.0 to 3.7]
Statistical Analysis 1: Comparison: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Response Rate Difference = 11.3, 95% CI 2-sided [7.2 to 15.3] — Difference = Upadacitinib 45 mg - Placebo

12. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 8
Description: The FACIT fatigue questionnaire was developed to assess fatigue associated with anemia. It consists of 13 fatigue-related questions. Each question is answered on a 5-point Likert scale: 0 (not at all); 1 (a little bit); 2 (somewhat); 3 (quite a bit); and 4 (very much). The total score ranges from 0 to 52, where higher scores represent less fatigue, and a positive change from Baseline indicates improvement.
Time Frame: Baseline (Week 0) to Week 8
Population: as for outcome 10
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Upadacitinib 45 mg | Placebo
Number analyzed (Participants) | 312 | 155
units on a scale | 9.4 [8.38 to 10.48] | 3.5 [2.02 to 4.92]
Statistical Analysis 1: Comparison: Upadacitinib 45 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed-effect model repeated measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 10, analysis 1]; LS Mean Difference = 6.0, 95% CI 2-sided [4.19 to 7.73], Standard Error of Mean 0.9 — Difference = Upadacitinib 45 mg - Placebo

ADVERSE EVENTS:
Time Frame: Part 1: From first dose of study drug up to 30 days after the last dose (up to 12 weeks) or until first dose of study drug in Part 2 or first dose of study drug in M14-234 (NCT02819635; maintenance study) or M14-533 (NCT03006068; long term extension). Part 2: From the first dose of study drug in Part 2 up to 30 days after last dose (up to 12 weeks) or until first dose of study drug in M14-234 (maintenance study) or the first dose date of study drug in M14-533 (long-term extension study).
Arm/Group | Part 1: Upadacitinib 45 mg | Part 1: Placebo | Part 2: Upadacitinib 45 mg / Upadacitinib 45 mg | Part 2: Placebo / Upadacitinib 45 mg
All-Cause Mortality (participants affected / at risk) | 0/344 | 0/177 | 0/68 | 0/116
Serious Adverse Events (participants affected / at risk) | 11/344 | 8/177 | 1/68 | 4/116
Other Adverse Events (participants affected / at risk) | 32/344 | 11/177 | 10/68 | 17/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Upadacitinib 45 mg (N=344) | Part 1: Placebo (N=177) | Part 2: Upadacitinib 45 mg / Upadacitinib 45 mg (N=68) | Part 2: Placebo / Upadacitinib 45 mg (N=116)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 4 (4) | 3 (3) | 1 (1) | 1 (1)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DENGUE FEVER (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENTEROCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ESCHERICHIA INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL STOMA NECROSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE PSYCHOSIS (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYODERMA GANGRENOSUM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Upadacitinib 45 mg (N=344) | Part 1: Placebo (N=177) | Part 2: Upadacitinib 45 mg / Upadacitinib 45 mg (N=68) | Part 2: Placebo / Upadacitinib 45 mg (N=116)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
HEADACHE (Nervous system disorders) | 8 (9) | 9 (10) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 24 (25) | 3 (3) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection

DOCUMENTS (2):
  • Study Protocol (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT03653026/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT03653026/SAP_001.pdf